CLINICAL TRIAL: NCT00567502
Title: A Non-Interventional, Post Authorisation Safety Study, to Continuously Monitor Safety and Pregnancy Outcomes in a Cohort of At-Risk Essential Thrombocythaemia (ET) Subjects Exposed to Xagrid Compared to Other Conventional Cytoreductive Treatments
Brief Title: Safety and Pregnancy Outcomes in Thrombocythemia Patients Exposed to XAGRID® (Anagrelide Hydrochloride) Compared to Other Treatments
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD422-401
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Thrombocythemia, Essential
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: XAGRID® (anagrelide hydrochloride)
- 2: Xagrid + Other cytoreductive
- 3: Other cytoreductive

SUMMARY:
This is an observational safety study being conducted in Europe comparing patients taking Xagrid to patients taking other cytoreductive treatments. The plan is to enrol at least 750 subjects taking Xagrid with up to 3000 subjects taking other cytoreductive therapies. The study will collect follow up data for 5 years for each patient enrolled that will focus on collecting data related to pre-defined events (PDEs) and Suspected Serious Adverse Reactions (SSARs).

ELIGIBILITY:
Inclusion Criteria:

* High risk ET patients
* Subjects who can give written informed consent.
* Subjects taking cytoreductive therapy

Exclusion Criteria:

* Contraindications listed by the product being used.
* Patient cannot be participating in another clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving cytoreductive therapy for the treatment of at-risk essential thrombocytopenia (ET).
Sampling Method: Probability Sample
Enrollment: 3647 (Actual)
Dates: Start 2005-05-31 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (164):
- Clinic of Haematology, Limassol, Cyprus
- Denmark (7):
  - Rigshospitalet, Copenhagen
  - SUS-Esbjerg Maematologisk afdelning, Esbjerg
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
  - Roskilde Sygehus, Roskilde
  - Vejle Sygehus, Vejle
  - Viborg Hospital, Viborg
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Jyvaskyla Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
- France (21):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier de Beauvais, Beauvais
  - Hopital Avicenne, Bobigny
  - Hopital de la Cavale Blanche, Brest
  - CHU Clemenceau, Caen
  - Hopital Henri Mondor, Créteil
  - Cabinet Medical, Dijon
  - Hopital Simone Veil, Eaubonne
  - CHU de Grenoble Hopital Albert Michallon, Grenoble
  - Centre Hospitalier de Lens, Lens
  - Hopital Saint Vincent de Paul, Lille
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - CHU de Limoges - Hopital Universitaire Dupuytren, Limoges
  - Centre Leon-Berard, Lyon
  - Hopital Nord, Marseille
  - C.H.U. de Nice Hopital de l Archet 1, Nice
  - Hopital Saint-Louis, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopital Hotel Dieu, Paris
  - Hopital Lariboisiere, Paris
  - Hopital Haut Leveque - CHU de Bordeaux, Pessac
- Germany (22):
  - Studienzentrum, Aschaffenburg
  - Praxis Dr. Heinrich, Dr. Brudler, Dr. Bangerter, Augsburg
  - Universitatsklinikum Koeln, Cologne
  - Praxis Schmitz and Steinmetz, Cologne
  - Hamatologisch-Onkologische Praxis, Dresden
  - Praxis Dr. Weniger und Dr. Bittrich, Erfurt
  - Onkologische Gemeinschaftspraxis, Frankfurt am Main
  - IORC GmbH, Hamburg
  - Hamburg
  - Internistische Praxis, Hornberg
  - Gemeinschaftspraxis fur Hamatologie und Internistische Onkologie, Magdeburg
  - Hamatologisch-Onkologische Praxis, Moers
  - Hamato-Onkologische Schwerpunktpraxis, Munich
  - Praxis Dr. Schick, München
  - Ambulante Chemotherapie, München
  - Hamatologisch-Onkologische Gemeinschaftspraxis, Münster
  - Praxis und Tagesklinik fur Internistische Onkologie, Recklinghausen
  - Caritasklinik St. Theresia, Saarbrücken
  - Schwerpunktpraxis fur Hamatologie und Internistische Onkologie, Saarbrücken
  - Universitatsklinik Ulm, Ulm
  - Hamatologie und Onkologie, Weiden
  - Praxis Dr. med. Yolanda Rodemer, Wilhelmshaven
- Greece (22):
  - 401 General Army Hospital, Athens
  - Henry Dunant Hospital, Athens
  - General Hospital of Athens G.Gennimatas, Athens
  - General Hospital of Athens Hippocratio, Athens
  - General Hospital of Athens Laiko, Athens
  - Laikon General Hospital of Athens, Athens
  - University Hospital of Athens Attikon, Athens
  - Hygeia Hospital, Athens
  - 3rd Hospital of IKA, Athens
  - General Hospital of Athens, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Athens ¿Attikon¿, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - Makarios Hospital, Nikiá
  - St. Andrews General Hospital of Patra, Pátrai
  - University Hospital of Patra, Pátrai
  - Piraeus
  - General Hospital of Thessaioniki, Thessaloniki
  - Ippokration Hospital D Clinic of Internal Medicine, Thessaloniki
  - Papageorgiou Hospital, Thessaloniki
- Midland Regional Hospital, Tullamore, Ireland
- Italy (41):
  - Ospedale Le Torrette, Ancona
  - Ospedale Arezzo, Arezzo
  - Ospedale Policlinico Consorziale, Bari
  - A.O. Spedali Civili di Brescia, Brescia
  - Presidio Ospedaliero Perrino, Brindisi
  - Ospedale Ferrarotto, Catania
  - Ospedale Civile, Civitanova Marche
  - Ospedale Santa Croce, Fano
  - Ospedale Careggi, Florence
  - Azienda Ospedaliera Ospedali Riuniti Foggia, Foggia
  - Ospedale S. Martino, Genova
  - Ospedale S.Martino, Genova
  - Ospedale San Martino, Genova
  - Ospedale San salvatore, L’Aquila
  - Ospedale Umberto I, Mestre
  - Policlinico, Modena
  - Azienda ospedaliera S. Gerardo, Monza
  - Ospedale A.Cardarelli, Napoli
  - Ospedale Cardarelli, Napoli
  - Universita Federico II, Napoli
  - Ospedale Maggiore della Carita, Novara
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Maggiore, Parma
  - IRCCS Policlinico S. Matteo, Pavia
  - Policlinico Monteluce, Perugia
  - Ospedale S. Salvatore, Pesaro
  - Ospedale Civile, Piacenza
  - Ospedale civile, Ragusa
  - Ospedale Santa Maria delle Croci, Ravenna
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - San camillo de Lellis, Rieti
  - Ospedale oncologico regionale, Rionero in Vulture
  - Policlinico Gemelli, Roma
  - Ospedale Nuova Regina Margherita, Rome
  - Ospedale Umberto I, Rome
  - Ospedale S.Spirito, Rome
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Padiglione ex-oncologico Ospedale S.Maria, Terni
  - Ospedale Luigi Gonzaga, Torino
  - Ospedale Molinette, Torino
  - Ospedale civile, Vigevano
- VU medical Center Amsterdam, Amsterdam, Netherlands
- Norway (4):
  - Sykehuset Ostfold, Fredrikstad
  - Universitetssykehuset Nord-Norge Hf, Tromsø
  - Trondheim
  - Akershus University Hospital, Viken
- Servico de Hematologia, Vila Nova de Gaia, Portugal
- Spain (16):
  - Hospital San Eloy, Barakaldo
  - Hospital del Mar, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Josep Trueta, Girona
  - Complexo Hospitalario Xeral Calde, Lugo
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital U. 12 de Octubre, Madrid
  - Hospital JM Morales Meseguer, Murcia
  - Hospital Clinico Universitario Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Clinico Universitario Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
- Sweden (12):
  - Falu Lasarett, Falun
  - Medicine Clinic, Gävle
  - Lanssjukhuset Ryhov, Jönköping
  - Ljungby Hospital Medical Clinic, Ljungby
  - University Hospital MAS, Malmo
  - University Hospital, Örebro
  - Sodersjukhuset - Medicinkliniken, Stockholm
  - Karolinska University Hospital, Stockholm
  - Lanssjukhuset Sundsvall - Harnosand, Sundsvall
  - Uddevalla Hospital, Uddevalla
  - Akademiska Hospital Uppsala, Uppsala
  - Centrallasarettet - Medicinavdelningen, Västerås
- United Kingdom (12):
  - Royal United Hospital, Bath
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Avon Haematology Unit BHOC, Bristol
  - Darlington Memorial Hospital, Darlington
  - Doncaster Royal Infirmary, Doncaster
  - Georgina Oncology Unit, Dudley
  - James Paget University Hospital, Great Yarmouth
  - Hull Royal Infirmary, Hull
  - Guy's and Thomas' NHS Foundation Trust, London
  - North Tyneside General Hospital, North Shields
  - Royal Shrewsbury Hospital, Shrewsbury

REFERENCES:
- [Derived] Birgegard G, Besses C, Griesshammer M, Gugliotta L, Harrison CN, Hamdani M, Wu J, Achenbach H, Kiladjian JJ. Treatment of essential thrombocythemia in Europe: a prospective long-term observational study of 3649 high-risk patients in the Evaluation of Anagrelide Efficacy and Long-term Safety study. Haematologica. 2018 Jan;103(1):51-60. doi: 10.3324/haematol.2017.174672. Epub 2017 Oct 27. PMID 29079600
- [Derived] Gugliotta L, Besses C, Griesshammer M, Harrison C, Kiladjian JJ, Coll R, Smith J, Abhyankar B, Birgegard G. Combination therapy of hydroxycarbamide with anagrelide in patients with essential thrombocythemia in the evaluation of Xagrid(R) efficacy and long-term safety study. Haematologica. 2014 Apr;99(4):679-87. doi: 10.3324/haematol.2012.083097. Epub 2013 Dec 13. PMID 24334294
- [Derived] Besses C, Kiladjian JJ, Griesshammer M, Gugliotta L, Harrison C, Coll R, Smith J, Abhyankar B, Birgegard G. Cytoreductive treatment patterns for essential thrombocythemia in Europe. Analysis of 3643 patients in the EXELS study. Leuk Res. 2013 Feb;37(2):162-8. doi: 10.1016/j.leukres.2012.11.004. Epub 2012 Nov 29. PMID 23199894
- [Derived] Kiladjian JJ, Besses C, Griesshammer M, Gugliotta L, Harrison C, Coll R, Smith J, Birgegard G. Efficacy and safety of cytoreductive therapies in patients with essential thrombocythaemia aged >80 years: an interim analysis of the EXELS study. Clin Drug Investig. 2013 Jan;33(1):55-63. doi: 10.1007/s40261-012-0042-0. PMID 23184668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were newly diagnosed (received no treatment at the time of study registration) or previously diagnosed with essential thrombocythemia (ET), receiving or continuing previous cytoreductive therapy were recruited in the study
Pre-assignment Details: Due to the non-interventional nature of the study, participants could be receiving XAGRID, XAGRID+Other (Cytoreductives), other (cytoreductives) and no essential thrombocythemia (ET) therapy. During the study participants could change the treatments.
Groups:
- XAGRID Only: Participants who received XAGRID at a dose and mode of administration managed as per investigator's discretion and the relevant Summary of Product Characteristics (SmPC) at the time of registering into the study for a 5 year observation period, during which participants were able to switch treatments per investigator's discretion
- XAGRID+Other (Cytoreductives): Participants who received XAGRID+Other (Cytoreductives) at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study for a 5 year observation period, during which participants were able to switch treatments per investigator's discretion. Other Cytoreductives included Hydroxyurea, Interferon- alpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
- Other (Cytoreductives): Participants who received other (Cytoreductives) at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study for a 5 year observation period, during which participants were able to switch treatments per investigator's discretion. Other Cytoreductives included Hydroxyurea, Interferon- alpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
- No Essential Thrombocythemia (ET) Therapy: Participants who were not receiving any cytoreductive treatment for at least 28 consecutive days at the time of registering into the study for a 5 year observation period, during which participants were able to switch treatments per investigator's discretion.
Period: Overall Study
Arm/Group | XAGRID Only | XAGRID+Other (Cytoreductives) | Other (Cytoreductives) | No Essential Thrombocythemia (ET) Therapy
Started | 804 | 141 | 2666 | 110
Initiated Treatment | 804 | 141 | 2666 | 38
Completed | 563 | 108 | 1758 | 23
Not Completed | 241 | 33 | 908 | 87
Not completed — Lost to Follow-up | 91 | 14 | 351 | 2
Not completed — Death | 65 | 16 | 360 | 5
Not completed — Other | 64 | 2 | 134 | 6
Not completed — Participant request | 12 | 1 | 33 | 1
Not completed — Sponsor request | 9 | 0 | 30 | 1
Not completed — Never Initiated Treatment | 0 | 0 | 0 | 72

BASELINE CHARACTERISTICS:
Population: First Treatment Safety Population included all participants who received at least 1 dose of cytoreductive treatment. Data of 2 participants were missing in the Other (Cytoreductives) treatment arm.
Groups:
- XAGRID+Other (Cytoreductives): Participants who received XAGRID along with Other cytoreductives drugs at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study for a 5 year observation period, during which participants were able to switch treatments per investigator's discretion. Other Cytoreductives included Hydroxyurea, Interferon- alpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
- Total: Total of all reporting groups
Arm/Group | XAGRID Only | XAGRID+Other (Cytoreductives) | Other (Cytoreductives) | No Essential Thrombocythemia (ET) Therapy | Total
Number analyzed (Participants) | 804 | 141 | 2664 | 38 | 3647
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (14.99) | 59.9 (13.74) | 67.4 (13.05) | 64.3 (14.26) | 64.4 (14.43)
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 65 years | 575 | 89 | 913 | 14 | 1591
  65-<75 years | 133 | 30 | 897 | 13 | 1073
  Greater than equal to (>=)75 years | 96 | 22 | 854 | 11 | 983
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 501 | 80 | 1632 | 25 | 2238
  Male | 303 | 61 | 1032 | 13 | 1409

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least One Pre-Defined Event (PDE), Deaths, Pregnancies
Description: Pre-defined events (PDEs) were evaluated whenever an event occurred and was defined by a panel of independent qualified physicians, blinded to cytoreductive therapy, validated all PDEs prior to analysis (Event Validation Panel). Non-PDE death only included deaths not recorded as outcome of another PDE.
Time Frame: Up to 5 years
Population: First Treatment Safety Population included participants who received cytoreductive therapy at registration. All events/data were allocated to the treatment that a participant was receiving at the time of the event/assessment.
Measure: Number; unit: percentage of participants
Groups:
- XAGRID Only: Participants who received XAGRID at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study or after switching from another treatment any time during the 5 year observation period.
- XAGRID+Other (Cytoreductives): Participants who received XAGRID+Other (Cytoreductives) at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study or after switching from another treatment any time during the 5 year observation period. Other Cytoreductives included Hydroxyurea, Interferon- alpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
- Other (Cytoreductives): Participants who received other (Cytoreductives) at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study or after switching from another treatment any time during the 5 year observation period. Other Cytoreductives included Hydroxyurea, Interferon- alpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
Arm/Group | XAGRID Only | XAGRID+Other (Cytoreductives) | Other (Cytoreductives)
Number analyzed (Participants) | 804 | 141 | 2666
percentage of participants
  Myocardial infarction | 1.0 | 0.0 | 1.5
  Angina | 0.7 | 0.0 | 0.7
  Congestive heart failure | 1.2 | 1.4 | 1.2
  Cardiomyopathy | 0.5 | 0.0 | 0.3
  Other cardiovascular symptoms | 5.8 | 8.5 | 3.2
  Stroke | 1.4 | 1.4 | 1.8
  Transient ischemic attack | 1.1 | 0.7 | 1.3
  Severe Mucocutaneous Disorders | 0.5 | 1.4 | 2.4
  Pulmonary hypertension | 0.5 | 0.0 | 0.2
  Pulmonary fibrosis/ Interstitial pneumonia | 0.1 | 0.0 | 0.3
  Venous thromboembolic events | 0.5 | 0.0 | 1.9
  Pancreatitis | 0.0 | 0.0 | 0.1
  Intermittent Claudication/ digital ischaemia | 0.7 | 0.7 | 0.6
  Transformations | 4.5 | 6.4 | 3.1
  Myelofibrosis | 3.5 | 5.0 | 1.1
  Myelodysplasia | 0.0 | 0.0 | 0.5
  Acute leukaemia | 0.2 | 1.4 | 1.0
  Other leukaemia | 0.6 | 0.0 | 0.5
  Other transformations | 0.1 | 0.0 | 0.1
  Major haemorrhagic events | 3.0 | 0.7 | 1.6
  Rhabdomyolysis/ myalgia | 0.2 | 0.0 | 0.1
  Non-haematological malignancy | 1.5 | 1.4 | 4.6
  Non-PDE death | 2.2 | 1.4 | 3.9
  Pregnancy | 0.5 | 0.0 | 0.5
  Thrombohaemorrhagic events | 8.1 | 3.5 | 8.5
  Major thrombotic events | 5.3 | 2.8 | 7.3
  Arterial events | 4.9 | 2.8 | 5.5

2. Secondary Outcome: Event Rate of Thrombohaemorrhagic Events
Description: Event Rate of Thrombohaemorrhagic Events was calculated by dividing number of participants with events by total patient-year exposure. The reporting unit is per 100 participant-years of treatment exposure. Thrombohaemorrhagic Events is a composite endpoint of the PDEs myocardial infarction, angina, stroke, transient ischaemic attack, venous thromboembolic events, intermittent claudication/digital ischaemia, and major haemorrhagic events.
Time Frame: Up to 5 years
Population: Overall Treatment Safety Population. As participant could switch between therapies a participant with an event could be allocated to more than one therapy group. Participants analyzed included who were exposed to the specific treatment any time during the study.
Measure: Number; unit: participants/100 participant-years
Arm/Group | XAGRID Only | XAGRID+Other (Cytoreductives) | Other (Cytoreductives) | No Essential Thrombocythemia (ET) Therapy
Number analyzed (Participants) | 1127 | 451 | 2909 | 645
participants/100 participant-years | 2.75 | 2.86 | 2.60 | 4.91

3. Secondary Outcome: Platelet Count
Time Frame: Baseline, Month 6,12,18, 24, 30, 36, 42, 48, 54, 60
Population: Overall Treatment Safety population, Here n = participants evaluable at specified time-points. As participant could switch between therapies a participant with an event could be allocated to more than one therapy group. Participants analyzed included who were exposed to the specific treatment any time during the study.
Measure: Mean (Standard Deviation); unit: 10^9 per Liter (10^9/L)
Groups:
- Other (Cytoreductives): Participants who received other (Cytoreductives) at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study or after switching from another treatment any time during the 5 year observation period.Other Cytoreductives included Hydroxyurea, Interferon- alpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
Arm/Group | XAGRID Only | XAGRID+Other (Cytoreductives) | Other (Cytoreductives) | No Essential Thrombocythemia (ET) Therapy
Number analyzed (Participants) | 1127 | 451 | 2909 | 645
10^9 per Liter (10^9/L)
  Baseline (n = 671, 120, 2279,136) | 486.90 (210.106) | 542.77 (250.440) | 471.29 (201.620) | 837.23 (377.104)
  Month 6 (n = 777, 145, 2469, 60) | 1093.73 (17634.779) | 521.44 (266.512) | 439.44 (153.766) | 545.30 (202.936)
  Month 12 (n= 739, 158, 2400, 81) | 969.61 (14404.677) | 516.66 (245.789) | 436.64 (154.958) | 501.46 (275.880)
  Month 18 (n= 706, 170, 2231, 86) | 1612.14 (22193.573) | 541.78 (706.564) | 432.99 (145.694) | 476.72 (245.450)
  Month 24 (n= 673, 181, 2106, 119) | 865.09 (11047.483) | 492.67 (194.534) | 1025.11 (15888.471) | 499.29 (249.164)
  Month 30 (n= 642, 183, 2001, 116) | 418.97 (159.129) | 467.37 (170.733) | 693.30 (8293.353) | 467.54 (255.641)
  Month 36 (n= 628, 167, 1917, 124) | 423.10 (153.278) | 1138.81 (8787.658) | 1221.09 (20612.960) | 462.06 (256.357)
  Month 42 (n= 597, 161, 1799, 138) | 831.62 (10257.081) | 466.83 (205.575) | 1898.48 (26724.419) | 463.52 (271.690)
  Month 48 (n= 581, 167, 1735, 131) | 2461.07 (28879.771) | 443.91 (173.453) | 1360.17 (20669.182) | 457.44 (250.165)
  Month 54 (n= 557, 164, 1644, 132) | 413.93 (145.601) | 447.17 (171.608) | 1771.77 (25187.992) | 408.41 (254.971)
  Month 60 (n = 523, 167, 1586, 144) | 1174.87 (17473.437) | 466.31 (193.689) | 1362.94 (19098.693) | 425.22 (268.377)

4. Secondary Outcome: Duration of Exposure for Each Essential Thrombocythemia (ET) Therapy
Description: Total duration for each participant = sum of [stop date - start date + 1] across all periods of time where the specific treatment was taken during the study, where start date = registration/consent date for treatments started before registration/consent date and/or stop date withdrawal/final date for treatments ongoing at the time of withdrawal/end of study. Where a participant has multiple records of the same therapy on the same day, the therapy is counted once for that day.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Groups:
- XAGRID Taken: Participants who received XAGRID from "Xagrid only" or "Xagrid+other (cytoreductives)" arm groups at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC at the time of registering into the study for a 5 year observation period.
- Other (Cytoreductives)-Hydroxyurea: Participants who received other (Cytoreductives)-Hydroxyurea at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other (Cytoreductives)-Interferon Alpha: Participants who received other (Cytoreductives)-Interferon Alpha at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other (Cytoreductives)-Pegylated Interferon: Participants who received other (Cytoreductives)-Pegylated Interferon at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other (Cytoreductives)-Busulphan: Participants who received other (Cytoreductives)-Busulphan at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other (Cytoreductives)-Pipobroman: Participants who received other (Cytoreductives)-Pipobroman at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other (Cytoreductives)-Sodium Phosphate P32: Participants who received other (Cytoreductives)-Sodium Phosphate P32 at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other (Cytoreductives)-Thromboreductin: Participants who received other (Cytoreductives)-Thromboreductin at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other: Participants who received other therapies at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
Arm/Group | XAGRID Taken | Other (Cytoreductives)-Hydroxyurea | Other (Cytoreductives)-Interferon Alpha | Other (Cytoreductives)-Pegylated Interferon | Other (Cytoreductives)-Busulphan | Other (Cytoreductives)-Pipobroman | Other (Cytoreductives)-Sodium Phosphate P32 | Other (Cytoreductives)-Thromboreductin | Other
Number analyzed (Participants) | 1300 | 2742 | 193 | 144 | 105 | 159 | 12 | 5 | 91
days | 1213.7 (687.83) | 1382.3 (609.33) | 933.3 (748.09) | 744.0 (660.93) | 510.2 (560.28) | 992.8 (690.80) | 39.7 (96.73) | 979.0 (859.27) | 446.3 (561.46)

5. Secondary Outcome: Cumulative Dose for Each Essential Thrombocythemia (ET) Therapy
Description: Since the study is observational nature, interpreting the table is difficult due to inconsistencies in reporting the units of the dose.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram (mg)
Groups:
- XAGRID Only: Participants who received XAGRID at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
Arm/Group | XAGRID Only | Other (Cytoreductives)-Hydroxyurea | Other (Cytoreductives)-Interferon Alpha | Other (Cytoreductives)-Pegylated Interferon | Other (Cytoreductives)-Busulphan | Other (Cytoreductives)-Pipobroman | Other (Cytoreductives)-Sodium Phosphate P32 | Other (Cytoreductives)-Thromboreductin | Other
Number analyzed (Participants) | 1162 | 2168 | 2 | 9 | 92 | 112 | 1 | 4 | 70
milligram (mg) | 29096.2 (291472.25) | 957751.4 (883174.77) | 3592.2 (5076.77) | 5103.1 (10730.47) | 7749.6 (56031.79) | 28612.7 (67374.96) | 2745.0 | 2140.0 (835.26) | 111639.7 (190370.57)

6. Primary Outcome: Number of Participants With Suspected Serious Adverse Reaction (SSAR) Events
Description: SSAR: serious adverse event (SAE) that was considered related to cytoreductive therapy. SAE: any untoward medical occurrence that at any dose resulted in death, life-threatening (at the time of the event), in-patient hospitalization/prolongation of existing hospitalization (elective hospitalizations/procedures for pre-existing conditions that had not worsened were excluded), resulted in persistent or significant disability/incapacity or congenital abnormality/birth defect. Relatedness (suspected/not suspected) to XAGRID or other cytoreductive theraphy was determined by the investigator. As for SSARs, it was important to consider whether the events were related to XAGRID or other cytoreductive therapy. A participant was included in Xagrid or other treatment group based on treatment exposure, participants received Xagrid + Other was counted both in Xagrid and other treatment group.
Time Frame: Up to 5 years
Population: Overall treatment safety population. All events/data were allocated to the treatment that a participant was receiving at the time of the event/assessment. Participants who had exposed to XAGRID (alone or in combination with other) was counted in Xagrid arm and those who had received other ET therapy in the "Other (Cytoreductives)".
Measure: Number; unit: participants
Groups:
- XAGRID: Participants who received XAGRID at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years.
- Other (Cytoreductives): Participants who received other (Cytoreductives) at a dose and mode of administration managed as per investigator's discretion and the relevant SmPC, was observed for 5 years. Other Cytoreductives included Hydroxyurea, Interferonalpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
Arm/Group | XAGRID | Other (Cytoreductives)
Number analyzed (Participants) | 1300 | 3069
participants | 37 | 70

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: SSARs [defined in outcome measure (OM) 2]= SAEs considered related to cytoreductive drug and only "XAGRID" and "Other" treatment groups were to be reported. SAEs and non-SAEs was not planned to be reported separately, therefore, reported under OM 1.
Groups:
- XAGRID: Participants who received XAGRID from "Xagrid only" or "Xagrid+other (cytoreductives)" arm groups (for serious adverse events) at a dose and mode of administration managed as per investigator's discretion and the relevant Summary of Product Characteristics (SmPC) at the time of registering into the study or after switching from another treatment (other adverse events) any time during the 5 year observation period.
- Other (Cytoreductives): Participants who received other (cytoreductives) from " other (cytoreductives" or "Xagrid+other (cytoreductives)" arm groups (for serious adverse events) at a dose and mode of administration managed as per investigator's discretion and the relevant Summary of Product Characteristics (SmPC) at the time of registering into the study or after switching from another treatment (other adverse events) any time during the 5 year observation period. Other Cytoreductives included Hydroxyurea, Interferon- alpha, Pegylated interferon, Busulphan, Pipobroman, Sodium phosphate P32.
Arm/Group | XAGRID | Other (Cytoreductives)
Serious Adverse Events (participants affected / at risk) | 37/1300 | 70/3069
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XAGRID (N=1300) | Other (Cytoreductives) (N=3069)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 9 (9)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure Congestive (Cardiac disorders) | 3 (3) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelodysplastic syndrome transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 4 (4)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Erythrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Results for other adverse events (excluding SAEs) was reported under OM 1 due to limitation in basic result's format, as SAEs and non-SAEs were not planned to be reported separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.